CLINICAL TRIAL: NCT03941509
Title: Stepped-wedge Cluster Randomised Controlled Trial to Increase Antibiotic Appropriateness in Residential Aged Care Facilities: a Nurse-led Bundled Antimicrobial Stewardship Intervention.
Brief Title: Nurse-led Antimicrobial Stewardship Intervention to Increase Antibiotic Appropriateness in Residential Aged Care Facilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Bupa Aged Care Australia (Unknown); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 591/18
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Antimicrobial Stewardship; Urinary Tract Infections; Respiratory Tract Infections; Skin and Soft Tissue Infections
MeSH Terms: conditions — Urinary Tract Infections; Respiratory Tract Infections; Soft Tissue Infections | interventions — Antimicrobial Stewardship

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design will see a staggered roll out of the intervention over 16 months. Each cluster of two facilities will commence in the control phase (2 months) and transition to the intervention phase until all facilities receive the intervention. A transition phase of 2 months between the control and intervention phase will occur to allow for education and integration of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): All facilities will receive usual care during the control phase of the trial.
- Antimicrobial stewardship (Experimental): Implementation of the nurse-led bundled antimicrobial stewardship intervention
  Interventions: Behavioral: Antimicrobial stewardship

INTERVENTIONS:
Behavioral: Antimicrobial stewardship — Education, guidelines, communication tools and audit and feedback
  Arms: Antimicrobial stewardship

SUMMARY:
The study will explore the impact of a nurse-led bundled antimicrobial stewardship intervention on the appropriateness of antimicrobial use in residential aged care facilities. The intervention will be assessed in a stepped-wedge cluster randomised controlled trial across 14 residential aged care facilities over an 18-month period.

DETAILED DESCRIPTION:
The study will explore the impact of a nurse-led bundled antimicrobial stewardship intervention on the appropriateness of antimicrobial use in residential aged care facilities (RACFs).

The antimicrobial stewardship intervention will include the following components:

1. Education

   * Focused on antimicrobial stewardship and appropriate antimicrobial use
   * Delivered face-to-face, via workbooks and fact sheets to aged care staff, general practitioners (GPs), pharmacists, and residents and families. Education will be delivered by the research coordinator.
2. Guidelines

   * Aged care-specific guidelines for the assessment and antimicrobial management of urinary tract infections, respiratory tract infections and skin and soft tissue infections.
   * Antimicrobial management recommendations including empirical oral therapy, doses and duration of therapy.
3. Communication

   * Documentation for the assessment and antimicrobial management of infections.
   * Nurse-led engagement with residents and families.
   * Newsletters and online updates to highlight evidence-based prescribing practice
4. Audit and feedback - Surveillance and feedback to prescribers on antimicrobial use and facility-level antimicrobial susceptibility data.

The intervention bundle will first be implemented and tested for feasibility and acceptability over a 3-month period in two RACFs in Victoria, Australia. This tailored intervention will then be assessed in a stepped-wedge cluster randomised controlled trial across 12 RACFs over an 16-month period.

A cluster of two facilities will each transition through three phases over the 16 month trial:

* Control phase: baseline data collection. Usual care at each facility.
* Transition phase: Delivery of education and integration of the intervention. No data collection.
* Intervention phase: implementation of the intervention and outcome data collection. Ongoing education to new and existing staff will be provided as required.

Following the 16-month trial, the refined intervention bundle will be implemented nationally across a network of RACFs.

ELIGIBILITY:
Inclusion Criteria:

Residents:

* All residents from 12 RACFs will have de-identified data collected including antimicrobial use, infection, hospitalisation and mortality.
* Residents or their guardians who provide informed consent to monthly biospecimen sampling and participation in one-on-one interviews or focus groups.

Health professionals:

- Health professionals (including aged care staff and GPs) who provide informed consent to participate in one-on-one interviews or focus groups.

Exclusion Criteria:

* Residents or their guardians who do not consent to biospecimen sampling and/or participation in interviews/focus groups.
* Health professionals who do not consent to participate in interviews/focus groups.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative proportion of residents prescribed a systemic antimicrobial | Assessed from commencement of the intervention at each facility until the conclusion of the trial at 16 months
Rate of total days of systemic antimicrobial therapy per 1,000 occupied bed days (OBD) | Assessed from commencement of the intervention at each facility until the conclusion of the trial at 16 months

SECONDARY OUTCOMES:
Number of courses of systemic antimicrobial therapy per 1,000 OBD. | Assessed from commencement of the intervention at each facility until the conclusion of the trial at 16 months
Proportion of appropriate antimicrobial use. | Assessed from commencement of the intervention at each facility until the conclusion of the trial at 16 months
  Antimicrobials will be considered to be appropriate if minimum criteria for their initiation are met according to guidelines by the Society of Healthcare Epidemiology of America.
Frequency of carriage of antimicrobial-resistant organisms | Assessed over a 12-month period during the trial (at least 2 months pre-intervention and 2 months post-intervention).
  Monthly biospecimen sampling will be collected from residents including nasal, faecal/rectal and wound specimens.
Rate of Clostridium Difficile infection | Assessed from commencement of the intervention at each facility until the conclusion of the trial at 16 months
Change in facility-level antimicrobial susceptibility profile | Assessed over a 12-month period during the trial (at least 2 months pre-intervention and 2 months post-intervention).
  Monthly biospecimen sampling will be collected from residents including nasal, faecal/rectal and wound specimens.
Incidence of resident transfer to hospital for infectious indications | Assessed from commencement of the intervention at each facility until the conclusion of the trial at 16 months
All-cause mortality | Assessed from commencement of the intervention at each facility until the conclusion of the trial at 16 months
Perceptions from stakeholders on quality and uptake of the intervention | Assessed at the conclusion of the trial at 16 months
  Semi-structured interviews conducted one-on-one or in moderated focus groups with stakeholders including aged care staff, GPs, residents and families.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Peleg, MBBS, PhD, FRACP, PhD, Principal Investigator — Monash University
Locations (1):
- Bupa residential aged care facilities, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Jokanovic N, Haines T, Cheng AC, Holt KE, Hilmer SN, Jeon YH, Stewardson AJ, Stuart RL, Spelman T, Peel TN, Peleg AY; START Trial Group. Multicentre stepped-wedge cluster randomised controlled trial of an antimicrobial stewardship programme in residential aged care: protocol for the START trial. BMJ Open. 2021 Mar 2;11(3):e046142. doi: 10.1136/bmjopen-2020-046142. PMID 33653766